CLINICAL TRIAL: NCT03640078
Title: Automated Reading of Anti-neutrophil Cytoplasmic Autoantibodies (ANCA), Indispensable Markers of Vasculitis
Brief Title: Automated Reading of Anti-neutrophil Cytoplasmic Autoantibodies, Indispensable Markers of Vasculitis
Acronym: ANCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-25
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Vasculitis patients The usual care of the sera will not be modified, only a phase of acquisition of the images will be added to the analysis of serum. (acquisition imaging)
  Interventions: Other: acquisition imaging

INTERVENTIONS:
Other: acquisition imaging — The usual care of the sera will not be modified, only a phase of acquisition of the images will be added to the analysis

SUMMARY:
Neutrophil cytoplasmic autoantibodies (ANCA) are essential serum markers in the diagnosis of vasculitis. Indirect immunofluorescence with microscope reading by two readers is the reference technique for their detection. In the AP-HM immunology laboratory we are looking for ANCAs in more than 7000 sera per year. The reading of the slides is time-consuming, dependent operator, and lacks standardization. In order to optimize these parameters, we propose the automation of ANCA reading by using a robotic platform developed in our laboratory and called ICARE (Immunofluorescence for Computed Antibodies Rational Evaluation). This microscopic imaging platform with automated reading is currently used in daily routine for the detection of anti-nuclear autoantibodies.

The objective of the project is to establish an algorithm allowing i) to automatically and reproducibly discriminate the positive ANCAs from the negative ANCAs and ii) to propose to the biologist a fluorescence aspect. The investigators will then validate this algorithm on 2000 consecutive routine samples sent to the laboratory for ANCA research.

The usual care will not be changed, only a phase of acquisition of the images will be added to the analysis.

The investigators expect to use this algorithm "ICARE / ANCA" in daily hospital routine and thus optimize the results with a real economic impact is 50% less reading time.

DETAILED DESCRIPTION:
Neutrophil cytoplasmic autoantibodies (ANCA) are essential serum markers in the diagnosis of vasculitis. Indirect immunofluorescence with microscope reading by two readers is the reference technique for their detection. In the AP-HM immunology laboratory we are looking for ANCAs in more than 7000 sera per year. The reading of the slides is time-consuming, dependent operator, and lacks standardization. In order to optimize these parameters, we propose the automation of ANCA reading by using a robotic platform developed in our laboratory and called ICARE (Immunofluorescence for Computed Antibodies Rational Evaluation). This microscopic imaging platform with automated reading is currently used in daily routine for the detection of anti-nuclear autoantibodies.

The objective of the project is to establish an algorithm allowing i) to automatically and reproducibly discriminate the positive ANCAs from the negative ANCAs and ii) to propose to the biologist a fluorescence aspect. The investigators will then validate this algorithm on 2000 consecutive routine samples sent to the laboratory for ANCA research.

The usual care will not be changed, only a phase of acquisition of the images will be added to the analysis.

The investigators expect to use this algorithm "ICARE / ANCA" in daily hospital routine and thus optimize the results with a real economic impact is 50% less reading time. . From a valorisation point of view, this project could be the subject of a publication in an international scientific journal, a patent filing and an exploitation with an industrial partner.

ELIGIBILITY:
Inclusion Criteria:

* Vasculitis patients having signed a consent

Exclusion Criteria:

* patients refusing to sign a consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
The number of positive ANCAs | 1 day
  The number of positive ANCAs detected in order to automatically and reliably discriminate against positive ANCAs from negative ANCAs

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaix de Marseille, Marseille, PACA, France